CLINICAL TRIAL: NCT04003909
Title: Effectiveness of Ultrasound-guided Erector Spinae Plane Block for Postoperative Pain Control in Hip Replacement Surgeries
Brief Title: Erector Spinae Plane Block for Postoperative Pain Control in Hip Replacement Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bassant M. Abdelhamid (Other)
Responsible Party: Sponsor-Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-147-2018
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Experimental): patients will have ultrasound guided ESP block before spinal anesthesia.
  Interventions: Procedure: ultrasound-guided Erector spinae plane block; Procedure: subarachonoid block
- Control group (Experimental): patients will have spinal Anesthesia without ESP block
  Interventions: Procedure: subarachonoid block

INTERVENTIONS:
Procedure: ultrasound-guided Erector spinae plane block — The patients will be in lateral position. A curvilinear array ultrasound probe will be placed in a transverse orientation at L4 level to identify the tip of the L4 transverse process. Local anesthetic infiltration of the superficial tissues, an echogenic 22-G block needle will be inserted inplane to the ultrasound beam in a cranial-to-caudal direction until contact made with the L4 transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle will be confirmed by injecting 0.5-1ml saline and seeing the fluid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total volume of 20ml bupivicaine 0.25% and 20 ml xylocaine 1% will be injected into the ESP on the affected side.
  Arms: ESP group
Procedure: subarachonoid block — Local anesthesia 2ml of lidocaine 2% will be applied intradermally to the needle entrance point. A 22-G block needle will be inserted, free cerebrospinal fluid flow will be observed and 20mg of hyperbaric bupivacaine 0.5% and 10μg of fentanyl will be injected for 30 seconds.

SUMMARY:
ESP block advantages include its simplicity, easy identifiable ultrasonographic landmarks and low risk for serious complications as injection is into tissue plane that is distant from pleura, major blood vessels and discrete nerves. Coupled with the fact that the erector spinae muscle and ESP extend down to the lumbar spine, ESP block was hypothesized to be performed at the level of L4. In a recent case report, ultrasound guided ESP block was successfully performed at L4 transverse process level for postoperative analgesia after total hip arthroplasty. However, confirmation of the efficacy of ESP block in hip replacement surgeries needed more investigation.

DETAILED DESCRIPTION:
This study will be performed in Cairo university hospital. Thirty adult patients of both sexes scheduled for hip replacement surgery under spinal anesthesia will be enrolled in the study.

All patients meeting the inclusion criteria will be randomly assigned to one of 2 groups, 15 per group:

Group E, ESP group (n=15): prior to surgical incision, patients will have ultrasound guided ESP block before spinal anesthesia.

Group C, Control group (n=15): prior to surgical incision, patients will have spinal Anesthesia without ESP block .

Patients will be randomly allocated by a computer-generated table into one of the study groups, the randomization sequence will be concealed in sealed opaque envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 40 to 65 years old
* Both sexes.
* ASA I-II.
* Undergo hip replacement surgery.
* Body mass index (BMI) from 18 to 35 kg/m2.

Exclusion Criteria:

* Patient refusal.
* Contraindication to regional anesthesia (bleeding disorder, use of any anticoagulants, local infection, etc. )
* BMI > 35.
* Known allergy to local anesthetics.
* ASA III-IV.
* Patients with difficulty in evaluating their level of pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperative
  Total morphine consumption in rescue boluses during 1st 24 hrs postoperatively.

SECONDARY OUTCOMES:
Visual analogue scale | 30 minutes,2,4, 6, 12, and 24 hours postoperative.
  Visual analogue scale at the following intervals:30 minutes,2,4, 6, 12, and 24 hours postoperative.
Duration of analgesia | 24 hours postoperative
  defined as the time interval from completion of local anesthetic administration till first need of rescue analgesic in the form of iv morphine
Incidence of complications | 24 hours
  Nerve injury, Hematoma formation, LA toxicity, Intravascular injection.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Rady, M.D., Principal Investigator — Cairo University; Amr abdelnasser, Study Director — Cairo University
Locations (1):
- Anesthesia Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth. 2018 Jun;47:5-6. doi: 10.1016/j.jclinane.2018.02.014. Epub 2018 Mar 6. No abstract available. PMID 29522966
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experiences of ultrasound-guided erector spinae plane block for thoracic vertebra surgery. J Clin Anesth. 2017 May;38:137. doi: 10.1016/j.jclinane.2016.12.028. Epub 2017 Feb 17. No abstract available. PMID 28372654 (Retraction: PMID 35396111 J Clin Anesth. 2022 Aug;79:110791)
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392